CLINICAL TRIAL: NCT04460872
Title: Locomotor Training With Testosterone to Promote Bone and Muscle Health
Brief Title: Locomotor Training With Testosterone to Promote Bone and Muscle Health After Spinal Cord Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: North Florida/South Georgia Veterans Health System (Other); Brooks Rehabilitation (Other); University of Florida (Other); VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Yarrow, Research Health Scientist, North Florida Foundation for Research and Education
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 649726
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injury; Spinal Cord Injuries; Trauma, Nervous System; Wounds and Injury; Central Nervous System Diseases; Spinal Cord Diseases; Gonadal Disorders; Endocrine System Diseases; Hypogonadism; Genital Diseases, Male; Spinal Cord Trauma; Injuries, Spinal Cord; Walking, Difficulty; Gait Disorders, Neurologic; Locomotion Disorder, Neurologic; Wounds and Injuries; Nervous System Diseases; Testosterone Deficiency; Androgen Deficiency; Hormone Deficiency
Keywords: Testosterone; Testosterone enanthate; Testosterone undecanoate; Testosterone 17 beta-cypionate; Methyltestosterone; Androgens; Hormones; Hormone Substitutes, and Hormone Antagonists; Physiologic Effects of Drugs; Pharmacologic Actions; Therapeutic Uses; Anabolic Agents; Testosterone Replacement Therapy; Dual Energy X ray Absorptiometry; Lean Tissue Mass; Body Composition; Muscle Strength; Muscle Mass; Bone Mineral Density; Adipose Tissue; Body Fat; Density, Bone; Bone Formation; Bone Resorption; Bone Density Conservation Agents; Magnetic Resonance Imaging; Walking; Ambulation; Locomotor; Locomotion; Treadmill; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Trauma, Nervous System; Wounds and Injuries; Central Nervous System Diseases; Spinal Cord Diseases; Gonadal Disorders; Endocrine System Diseases; Hypogonadism; Genital Diseases, Male; Mobility Limitation; Gait Disorders, Neurologic; Nervous System Diseases; Bone Resorption | interventions — testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- testosterone enanthate (Experimental): Testosterone enanthate via i.m. injection (100 mg/week)
  Interventions: Drug: Testosterone Enanthate
- locomotor training, testosterone enanthate (Experimental): Treadmill and overground walking training and testosterone enanthate via i.m. injection (100 mg/week)
  Interventions: Drug: Testosterone Enanthate; Behavioral: Locomotor Training
- non-interventional control (No Intervention): Non-interventional control group

INTERVENTIONS:
Drug: Testosterone Enanthate — Subjects receive testosterone (100 mg/week) by intramuscular injection
  Other Names: delatestryl
  Arms: locomotor training, testosterone enanthate; testosterone enanthate
Behavioral: Locomotor Training — Subjects receive locomotor training (4 sessions/week for 2-3 months)
  Other Names: Treadmill training and overground walking
  Arms: locomotor training, testosterone enanthate

SUMMARY:
This pilot study will determine the feasibility of implementing a combinatory rehabilitation strategy involving testosterone replacement therapy (TRT) with locomotor training (LT; walking on a treadmill with assistance and overground walking) in men with testosterone deficiency and walking dysfunction after incomplete or complete spinal cord injury. The investigators hypothesize that LT+TRT treatment will improve muscle size and bone mineral density in men with low T and ambulatory dysfunction after incomplete or complete SCI, along with muscle fundtion and walking recovery in men with T low and ambulatory dysfunction ater incomplete SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) produces bone, muscle, and neural impairments that increase fracture risk and impede recovery of physical function. Locomotor training (LT) increases muscle size and promotes recovery of muscle function and walking in some persons with incomplete SCI. It is unknown if testosterone replacement therapy (TRT) improves these factors in men who have walking dysfunction and low testosterone after incomplete SCI. In addition, the combined effects of LT plus TRT remain unknown in men with incomplete SCI.

For this pilot study, men with incomplete SCI involving spinal level L1 or above for >60-days or complete SCI involving spinal levels T2-L1 for >60-days, with upper motor neuron signs, who have low testosterone and walking dysfunction will receive 6-months of TRT alone or TRT with LT. TRT injections will be given weekly. LT will involve 35 sessions of treadmill walking with assistance and overground walking (4 sessions per week) during the initial 2-3 months of TRT. Participants will be assessed at study entry and at 1-6 month intervals thereafter. Testing will include measurements such as a magnetic resonance imaging (MRI) scans, dual energy x-ray absorptiometry (DEXA) scan, and muscle performance and walking tests. Participants will also undergo safety tests, including physical exams, electrocardiogram (ECG), prostate digital rectal exam, and blood tests to assess hematocrit, liver enzymes (AST and ALT), prostate specific antigen (PSA), and other health markers. The treatment groups will be compared with a non-treatment control group comprised of men with incomplete or complete SCI who receive no treatment. Participants enrolled in the non-treatment control group will undergo the same tests described above.

ELIGIBILITY:
Inclusion Criteria:

* Men >18 years of age
* Diagnosis of an incomplete SCI involving spinal segments L1 or above or a clinically complete SCI involving spinal segments T2-L1, with upper motor neuron injury signs (i.e., spasticity, hypertonicity) for >60-days
* Low serum total testosterone (<300 ng/dL), bioavailable testosterone (<110 ng/dL), or free testosterone (<46 pg/mL or <4.6 ng/dL)
* Presence of one or more sign or symptom that may be related to low testosterone, including: loss of body hair or reduced shaving, very small testes (<6 mL), reduced sexual desire (libido) and activity, decreased spontaneous erections (e.g., morning erections) or erectile dysfunction, breast discomfort or gynecomastia, height loss, low-trauma fracture, or low BMD, hot flushes or sweats, decreased energy, motivation, initiative, or self-confidence, fatigue or irritability, feeling sad or blue, having a depressed mood, or having a persistent low-grade depressive disorder, poor concentration or memory, sleep disturbances or increased sleepiness, mild unexplained anemia (normochromic or normocytic), reduced muscle bulk, strength, or physical performance, Increased body fat or body mass index, any other sign or symptom commonly associated with low testosterone
* Locomotor dysfunction, definted as self-selected walking pace ≤1.0 m/s on a 10mWT, either with or without gait devices or braces and with or without assistance, or as self-selected walking pace >1.0 m/s with reliance on a gait device or brace or with highly compensated movement impairments, as identified by a trained observer.
* Diagnosis of first time SCI including etiology from trauma, vascular, or orthopedic pathology
* Medically-stable condition that is asymptomatic for conditions that will interfere with the study participation
* Willingness to administer TRT as instructed by the study staff and to abide by study protocol
* Documented approval from the study physician verifying medical status

Exclusion Criteria:

* Currently participating in another research protocol that may influence study outcomes.
* Mental state that precludes understanding the study protocol.
* Life expectancy <12-months.
* History of or current congenital SCI (e.g., Chiari malformation, myelomeningocele, intraspinal neoplasm, Frederich's ataxis) or other degenerative spinal disorder (e.g., spinocerebellar degeneration) that may complicate study procedures
* Multiple sclerosis, amyotrophic lateral sclerosis, or other neurologic impairment or injury
* Current prostate, breast, or other organ cancer or a history of prostate or breast cancer
* Any other diagnosed or treated cancer within the past 24-months, with the exceptions of basal or squamous cell carcinoma of the skin that has been successfully treated
* Serum prostate-specific antigen (PSA) >3.0 ng/mL [men treated with 5-alpha reductase inhibitors (e.g., finasteride or dutasteride) are eligible to participate if PSA values are ≤1.5 ng/mL]
* Prostate nodule or induration noted on digital rectal exam (DRE) during screening that tests positive for prostate cancer
* Currently seeking fertility or expected during the duration of the study
* Gynecomastia
* Hematocrit (HCT) >49%
* Any major cardiovascular (CV) event within the last 12-months (defined as a history of acute myocardial infarction, any cardiac revascularization procedure including angioplasty, stenting, or coronary artery bypass grafting, revascularization of the carotid or middle cerebral artery or procedures to treat critical limb ischemia, or hospitalization due to unstable angina, transient ischemic attack, stroke, or peripheral vascular disease)
* Angina that is not controlled on a current medical regimen (Canadian class II, III, or IV)
* Poorly compensated congestive heart failure (NYHA class III or IV)
* Poorly controlled hypertension (consistently measured systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg), while on medications
* Poorly controlled arrhythmia of any type
* Severe valvular heart disease
* Baseline electrocardiogram (ECG) findings such as left bundle branch block or marked ECG abnormalities that would preclude serial screening evaluations for occult ischemic events
* History of unprovoked deep venous thrombosis (DVT), unprovoked pulmonary embolism, history of recurrent DVT or known thrombophilia
* LDL cholesterol >160 mg/dL with history of any major CV event, defined above, within the last 12-months
* Major non-CV surgery (e.g., major abdominal or thoracic procedure) within 90-days prior to screening and/or a major surgery scheduled at the time of screening
* Liver enzymes (AST or ALT) >1.5 times the normal upper limit
* Severe or end-stage chronic kidney disease documented by estimated glomerular filtration rate (eGFR) <30 mL/min
* Diagnosed, but untreated severe obstructive sleep apnea
* Lower extremity fracture in the last 12-months (exclusion criterion for participation in LT+TRT group only)
* Femoral neck, total hip, or lumbar spine t-score below -2.5 or distal femur BMD <0.70 g/cm2, assessed via DEXA at screening (exclusion criterion for participation in LT+TRT group only)
* Current anticoagulant therapy (contraindication for i.m. injections)
* Use of any of the following pharmacologic agents in the previous 90-days: any TRT formulation, any compounded or over-the-counter androgenic hormones or androgen precursors, clomiphene, aromatase inhibitors, anti-estrogen or estrogen treatment, or growth hormone
* Use of anti-resorptive or bone anabolic drug therapy in the previous 180-days
* Acute use (>5-days) of any opioids (e.g., oxycodone, hydrocodone, etc) or systemic glucocorticoids >7.5 mg/d prednisone equivalent (e.g., hydrocortisone 30 mg, methylprednisolone 6 mg, or dexamethasone 1.2 mg) within 1-week before screening visit, except men who are taking these medications for a chronic condition and are anticipated to continue treatment for the study duration
* Known allergy to any component of the TRT formulation (e.g., sesame oil or cottonseed oil)
* Any other condition, therapy, lab abnormality, medical or psychiatric conditions, or reason that might pose a risk to the participant, make participation not in the person's best interest, confound the study results (e.g., inability to comply with study requirements), make the participant unsuitable to receive study intervention, or interfere with the person's ability to participate for the entire study duration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male
Enrollment: 21 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
change in thigh muscle cross-sectional area | baseline, 3 months, 6 months
  change in thigh muscle cross-sectional area assessed via MRI
change in 6 min walk test (6MWT) | baseline, 1 month, 3 months, 6 months
  change in distance covered on 6MWT
change in distal femur bone mineral density | baseline, 3 months, 6 months
  change in distal femur bone mineral density (BMD) assessed via DEXA

SECONDARY OUTCOMES:
change in knee extensor peak torque | baseline, 3 months, 6 months
  change in knee extensor peak torque assessed via dynamometry
change in 10m walk test (10mWT) | baseline, 1 month, 3 months, 6 months
  change in time to complete 10mWT
change in bone resorption marker | baseline, 3 months, 6 months
  change in circulating bone resorption marker
change in bone formation marker | baseline, 3 months, 6 months
  change in circulating bone formation marker

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Yarrow, PhD, Study Director — North Florida/South Georgia Veterans Health System; Dana M Otzel, Phd, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (2):
- United States (2):
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - Brooks Rehabilitation, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.
Time Frame: Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.
Access Criteria: Data will be shared according to the requirements described by the Department of Veterans Affairs, Office of Research & Development.